CLINICAL TRIAL: NCT06289569
Title: Home Tele Rehabilitation Therapy for Vascular Dementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Timea Hodics, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00037243
Record Dates: First submitted 2024-02-21; First posted 2024-03-04 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Dementia, Vascular; Stroke Sequelae
MeSH Terms: conditions — Dementia, Vascular

STUDY DESIGN:
Masking Description: Self-report measures will be not blinded, assessors will be blinded to treatment phase (SOC or telerehabilitation)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele Rehabilitation (Experimental): Telerehabilitation therapy Occupational therapist prescribed hand/arm exercises will continue for 90 minutes per day with adequate rest periods for 4 weeks, followed by telerehabilitation with the application for 4 weeks, when subjects will perform the tasks at home with the guidance of the treatment app. Detailed records of each subject's motor tasks, number of repetition and level of performance will be kept. Treatment will be performed Monday-Friday for approximately 4 weeks. Treatment times can be broken up into multiple treatment periods to accommodate patient and caregiver preferences.
  Interventions: Other: Home telerehabilitation therapy

INTERVENTIONS:
Other: Home telerehabilitation therapy — Occupational therapist prescribed hand/arm exercises will be assigned to patients. Records of each subject's motor tasks, number of repetition and level of performance will be kept. Standard of care home therapy will be performed Monday-Friday for approximately 4 weeks, followed by 4 weeks of application-driven home teletherapy. It is expected that approximately 20 treatments will be finished in 4weeks, however the amount of therapy completed will be recorded to accommodate patients' schedules. Treatment times can be broken up into multiple treatment periods to accommodate patient and caregiver preferences.

SUMMARY:
To determine whether the home telerehabilitation therapy is feasible and lessens caregiver burden in chronic stroke patients with and without vascular dementia (VaD)

DETAILED DESCRIPTION:
This is a controlled evaluator masked parallel study of chronic (>6mo from stroke onset) ischemic or hemorrhagic stroke patients diagnosed with and without vascular dementia to test the feasibility and effect of remote rehabilitation therapy targeting the weaker arm compared to usual care. All patients will undergo baseline evaluation, then usual care for 1 month followed by a remote telerehabilitation treatment for one month, followed by an evaluation 1 month after the completion of treatment.

Research procedures:

Subject Recruitment/Screening: Participants will be recruited from the PI's stroke recovery specialty clinic, and the Houston Methodist Hospital system by flyers and educating clinicians about the proposed study and the patient requirements. Prospective participants may also be identified through mining electronic medical records for ICD-9 and ICD-10 codes for stroke and hemiparesis for potentially eligible participants. Participants that appear to meet eligibility criteria based on the phone screening and medical record review will be invited to participate in an in-person screening session to ensure that they met the full inclusion criteria prior to being enrolled in the study.

Throughout all study visits subjects will be monitored for safety, comfort and any adverse events by trained study staff.

Initial Evaluation/Dependent Measures: The subject's initial evaluation will include questionnaires and impairment and functional scales. We will record demographic information, brain imaging, stroke history and medical history and medications from electronic medical records. We will store the deidentified brain imaging in XNAT under a study identifier on the secure server available at HMH.

Intervention:

All subjects will perform first their conventional home rehabilitation for 4 weeks followed by telerehabilitation therapy.

Occupational therapist prescribed hand/arm exercises will continue for 90 minutes per day with adequate rest periods.

Self-report measures will not be blinded. The investigator who determines the primary outcome measure will not be aware of treatment phase completed or prior performance (single-blind study design). Each treatment session will be expected to take approximately 1 hour 45 minute with prior setup and stretching. Treatment times can be broken up into multiple treatment periods to accommodate patient and caregiver preferences.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic ischemic or hemorrhagic stroke verified by computerized axial tomography or magnetic resonance imaging
* at least 6 months post stroke
* At least some active movement in the affected upper extremity (MRS 1 or more in shoulder elbow or wrist)
* Ability to provide informed consent, or LAR able to provide consent
* Expressed willingness to comply with all study procedures and attend all study-related visits for both the patient and at least one caregiver.
* Age ≥ 18.
* Ability to follow one-step commands.
* Community-dwelling with transportation to evaluation sessions.
* Ability to operate the therapy system with minimal assistance, including sufficient corrected vision to perceive objects from a distance of 5 feet.
* Modified Ashworth Scale Score 3 or less in the involved upper extremity
* Passive range of motion within functional ranges at the shoulder, elbow, wrist and hand

Exclusion Criteria:

* Patients with history of severe alcohol or drug abuse, psychiatric illnesses like severe depression, poor motivational capacity, or severe language disturbances, particularly of receptive nature or with serious cognitive deficits (defined as unable to follow study instructions even with help from caregiver).
* Patients with bilateral paresis, or weakness or sensory damage due to peripheral causes (e.g. peripheral nerve injury, muscle or orthopedic injury etc.)
* Patients with severe uncontrolled medical problems that would render intensive rehabilitation unfeasible or unsafe (e.g. cardiovascular disease, unstable cardiac arrhythmia, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, or a deteriorated condition due to age, epilepsy or others).
* Concurrent participation in other experimental upper extremity rehabilitation trials that would interfere with results.
* Non-English-speaking individuals will only be eligible if they can provide the appropriate translator for all the sessions of the study as no funding is available to pay for such services. However, we plan to include them once funding has been secured in the subsequent larger trial.
* Pregnancy
* Prisoners

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-14 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Burden Scale for Family Caregivers | 3-4 months
  Burden Scale for Family Caregivers BSFC-s[8] Subjective caregiver burden 10-item short version of the questionnaire.
Adverse events | 3-4 months
  Prospective record of adverse events including dropouts

SECONDARY OUTCOMES:
Fugl-Meyer Upper extremity assessment | 3-4 months
  The uFM test measures both proximal and distal upper extremity movements. Intratester and intertester reliability and validity of the Fugl-Meyer scale is well established in stroke patients. A score ranges 0-66, higher scores are better.
Wolf Motor Function Test (WMFT) | 3-4 months
  The WMFT is a time-based method to evaluate upper extremity performance of 17 tasks while providing insight into joint-specific and total limb movements. Lower time scores mean better motor function.

OTHER OUTCOMES:
Exercise log | 3-4 months
  Exercise log to record amount of use.
Stroke Impact Scale | 3-4 months
  Stroke Impact Scale (SIS) self-report questionnaire. Scale ranges 0-100, higher score means better recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Timea Hodics, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No